CLINICAL TRIAL: NCT04559607
Title: TACE Combined With Camrelizumab and Apatinib Versus TACE in Intermediate and Advanced Hepatocelluar Carcinoma: a Randomized, Open-label, Multi-center Clinical Trials
Brief Title: TACE Combined With Camrelizumab and Apatinib in Intermediate and Advanced Hepatocelluar Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Chief physician, Zhongda Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-HCC-II-005
Record Dates: First submitted 2020-09-09; First posted 2020-09-23 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: TACE+Camrelizumab+Apatinib (Experimental): Camrelizumab (iv. infusion of 200 mg); Apatinib (po. administration of 250 mg); TACE
  Interventions: Drug: Camrelizumab; Device: TACE; Drug: Apatinib
- Control group: TACE (Active Comparator): TACE
  Interventions: Device: TACE

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab: 200mg, iv, Q3W
  Arms: Experimental group: TACE+Camrelizumab+Apatinib
Device: TACE — TACE if necessary
Drug: Apatinib — Apatinib: 250m, po, QD
  Arms: Experimental group: TACE+Camrelizumab+Apatinib

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of TACE in combination with Camrelizumab and Apatinib versus TACE in patients with intermediate- and advanced HCC.

DETAILED DESCRIPTION:
This is a multicentric open-labal trial to evaluate the efficacy and safety of transarterial chemoembolization (TACE) in combination with Camrelizumab and Apatinib versus TACE in patients with intermediate- and advanced hepatocellular carcinoma (HCC). The primary hypotheses is that TACE in combination with Camrelizumab and Apatinib is superior to TACE alone with respect to progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of HCC confirmed by radiology, histology, or cytology

  -≥18 years
* China liver cancer staging: Ib-IIIa
* Child-Pugh score ≤6 point
* Previous TACE treatment(≤2 times) is permitted
* Adequate organ and marrow function

Exclusion Criteria:

* Participants who had another previous or current malignant tumor, except for early-stage cancer with low risk of recurrence or a malignant tumor curatively treated >5 years prior to enrolment with no recurrence
* Participants who have severe allergy to iodine, and unable to receive TACE
* Participants who have undergone a liver transplant or allogeneic bone marrow transplantation, or those who are in the waiting list for liver or bone marrow transplantation
* Participants who had congenital or acquired immune deficiency, such as HIV infection
* Participants who had a history of gastrointestinal bleeding within 6 months prior to randomization or a definite tendency of gastrointestinal bleeding
* Participants who had undergone arterial thromboembolism within 6 months prior to randomization or a definite tendency of gastrointestinal bleeding, such as cerebrovascular accident, ≥ CTCAE grade 3 deep vein thrombosis and pulmonary embolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) by investigator | Up to ~2 years
  PFS is defined as the time from randomization to progression or death from any cause. Progression in this trial was determined as untreatable (UnTACEable) progression, defined as the inability of a patients to further receive or benefit from TACE for reasons. Progression in this trial also included progression that met the JSH criteria for TACE failure/refractoriness.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to ~4 years
  OS is defined as the time from randomization to death from any cause.
PFS by investigator according to modified Response Evaluation Criteria in Solid Tumors (mRECIST) | Up to ~2 years
  PFS by investigator according to modified Response Evaluation Criteria in Solid Tumors (mRECIST)
Time to untreatable (unTACEable) progression (TTUP) by investigator | Up to ~2 years
  TTUP is defined as the time from randomization to Child-Pugh grade C, intrahepatic tumor progression (>50% increase vs baseline), MVI or EHS (diameter>10 mm), and met the JSH criteria for TACE failure/refractoriness.

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, Doctor, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No